CLINICAL TRIAL: NCT04398511
Title: The Effect of Lactobacillus Brevis CD2 on Traumatic Oral Lesions Induced by Fixed Orthodontic Appliance: a Randomized Clinical Trial
Brief Title: L Brevis for Traumatic Oral Lesions in Orthodontic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade de Passo Fundo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Fernando Fornari, Professor, Universidade de Passo Fundo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: University of Passo Fundo
Record Dates: First submitted 2020-05-16; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Orthodontic Appliance Complication; Oral Mucositis; Bacterium; Agent
Keywords: Fixed orthodontic appliance; Lactobacillus brevis CD2; Oral pain; Traumatic oral lesions
MeSH Terms: conditions — Stomatitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients were treated with identical lozenges containing probiotic or placebo. The treatments were revealed only after statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L brevis (Experimental): Lactobacillus brevis CD2 in lozenges containing 4 billion CFU. Patients used a lozenge 15 min after breakfast, lunch and dinner, during 21 days, starting in the day of installation of the orthodontic appliance.
  Interventions: Drug: L brevis
- Placebo (Placebo Comparator): Placebo in lozenges, identical to those of L brevis. Patients used a lozenge 15 min after breakfast, lunch and dinner, during 21 days, starting in the day of installation of the orthodontic appliance.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L brevis — Lactobacillus brevis CD2 lozenges (4 billion CFU) after breakfast, lunch and dinner for 21 days.
  Other Names: Oral probiotic
  Arms: L brevis
Drug: Placebo — Placebo lozenges after breakfast, lunch and dinner for 21 days.
  Arms: Placebo

SUMMARY:
Introduction: Traumatic oral lesions are common in the beginning of the orthodontic treatment, and pathogenic oral bacteria might be involved. We tested whether the probiotic Lactobacillus brevis CD2 (L brevis) is benefic in this condition. Methods: In a double-blind clinical trial, 20 patients were randomized to 21 days course of lozenges containing L brevis CD2 (4 billion colony-forming units after breakfast, lunch and dinner) or placebo, starting on the day of installation of the fixed orthodontic appliance. Main outcomes were days without oral lesions and oral pain score [ranging between 0 (no pain) and 10 (maximum)]. Oral health related quality of life was measured by OHIP-14 before and after treatments.

DETAILED DESCRIPTION:
Study protocol After signing the informed consent form, the patients underwent an oral examination and answered about clinical information, oral pain scale, and the OHIP-14 questionnaire. The pain scale was graded between 0 (no pain) and 10 (maximum), Likert standard. There was also a drawing for the distribution of coded treatments, through a number taken by the patient from a manila envelope. After the orthodontic appliance installation session, each patient was instructed to use the coded treatment for the next 21 days, two gums after breakfast, after lunch and after dinner, totalizing 12 billion UFC of L brevis or placebo per day. The patient was provided with a diary to note the daily appearance of lesions and their evolution during the 21-day period, as well as the occurrence of any new symptoms (potential adverse effect), in addition to proof of the commitment assumed by the use of the tablets. After 21 days, each patient was reexamined by the author of the study, who collected the diaries and obtained information regarding the oral examination, oral pain scale, data on adherence to treatment and self-completion of the OHIP-14.

Statistical analysis Quantitative data are described with mean and standard deviation (or standard error of the mean) or median and range, while qualitative data are displayed with absolute and relative frequencies. Student's t-test was used for comparison of quantitative data between groups, Wilcoxon-Mann-Whitney (WMW) test being employed when the assumptions for that test were not met. Exact chi-square and Fisher´s exact test (FET) were used for categorical data. Treatment effect on OHIP-14 was analyzed using a Generalize Estimating Equations (GEE) model with Poisson distribution and log link, the predictors being treatment, time (beginning and end of treatment) and interaction treatment*time. The analyses were performed with softwares GraphPrism version 4.0 and SPSS® (IBM SPSS statistics v18). Sample size was estimated using WinPEPI v11.65. The P value indicative of significance was < 0.05. Because the final outcome was prevention or mitigation (not maintenance or augmentation) of undesirable symptoms, one-tailed tests were used for comparisons between groups respect to days without oral lesions, oral pain and OHIP-14 scores.

ELIGIBILITY:
Inclusion Criteria:

* need for orthodontic treatment with fixed appliance

Exclusion Criteria:

* Oral lesions
* Uncompensated systemic diseases
* Regular use of corticoids, antibiotics, immuno regulators and antidepressive agents

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Number of days without traumatic oral lesions | First 21 days after appliance installation
  Oral lesions (ulcers) due to fixed orthodontic appliance
Oral pain scale | First 21 days after appliance installation
  Oral pain score measured by Likert scale between 0 (no pain) and 10 (maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fornari, Prof., Principal Investigator — University of Passo Fundo
Locations (1):
- Post-Graduate Program in Dentistry, Passo Fundo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rennick LA, Campbell PM, Naidu A, Taylor RW, Buschang PH. Effectiveness of a novel topical powder on the treatment of traumatic oral ulcers in orthodontic patients: A randomized controlled trial. Angle Orthod. 2016 May;86(3):351-7. doi: 10.2319/050415-303.1. Epub 2015 Sep 24. PMID 26401826
- [Background] Kluemper GT, Hiser DG, Rayens MK, Jay MJ. Efficacy of a wax containing benzocaine in the relief of oral mucosal pain caused by orthodontic appliances. Am J Orthod Dentofacial Orthop. 2002 Oct;122(4):359-65. doi: 10.1067/mod.2002.126405. PMID 12411880
- [Background] Bagatin CR, Andrucioli MCD, Ferreira JTL, Matsumoto MAN, da Silva RAB, da Silva LAB, Romano FL, Nelson-Filho P. Biofilm formation in Haas palatal expanders with and without use of an antimicrobial agent: an in situ study. Microsc Res Tech. 2017 May;80(5):471-477. doi: 10.1002/jemt.22817. Epub 2016 Dec 9. PMID 27935660
- [Background] Gizani S, Petsi G, Twetman S, Caroni C, Makou M, Papagianoulis L. Effect of the probiotic bacterium Lactobacillus reuteri on white spot lesion development in orthodontic patients. Eur J Orthod. 2016 Feb;38(1):85-89. doi: 10.1093/ejo/cjv015. Epub 2015 Apr 3. PMID 25840585
- [Background] Anusha RL, Umar D, Basheer B, Baroudi K. The magic of magic bugs in oral cavity: Probiotics. J Adv Pharm Technol Res. 2015 Apr-Jun;6(2):43-7. doi: 10.4103/2231-4040.154526. PMID 25878972
- [Background] Haukioja A. Probiotics and oral health. Eur J Dent. 2010 Jul;4(3):348-55. PMID 20613927
- [Background] Rastogi P, Saini H, Dixit J, Singhal R. Probiotics and oral health. Natl J Maxillofac Surg. 2011 Jan;2(1):6-9. doi: 10.4103/0975-5950.85845. PMID 22442601
- [Background] Riccia DN, Bizzini F, Perilli MG, Polimeni A, Trinchieri V, Amicosante G, Cifone MG. Anti-inflammatory effects of Lactobacillus brevis (CD2) on periodontal disease. Oral Dis. 2007 Jul;13(4):376-85. doi: 10.1111/j.1601-0825.2006.01291.x. PMID 17577323
- [Background] Sharma A, Rath GK, Chaudhary SP, Thakar A, Mohanti BK, Bahadur S. Lactobacillus brevis CD2 lozenges reduce radiation- and chemotherapy-induced mucositis in patients with head and neck cancer: a randomized double-blind placebo-controlled study. Eur J Cancer. 2012 Apr;48(6):875-81. doi: 10.1016/j.ejca.2011.06.010. Epub 2011 Jul 6. PMID 21741230
- [Background] Sharma A, Tilak T, Bakhshi S, Raina V, Kumar L, Chaudhary S, Sahoo R, Gupta R, Thulkar S. Lactobacillus brevis CD2 lozenges prevent oral mucositis in patients undergoing high dose chemotherapy followed by haematopoietic stem cell transplantation. ESMO Open. 2017 Feb 13;1(6):e000138. doi: 10.1136/esmoopen-2016-000138. eCollection 2016. PMID 28848667
- [Background] Lee JK, Kim SJ, Ko SH, Ouwehand AC, Ma DS. Modulation of the host response by probiotic Lactobacillus brevis CD2 in experimental gingivitis. Oral Dis. 2015 Sep;21(6):705-12. doi: 10.1111/odi.12332. Epub 2015 Apr 20. PMID 25720615